CLINICAL TRIAL: NCT06502951
Title: Upper Cervical Spine Manipulation and Dry Needling Versus Conventional Physical Therapy in Patients With Cervicogenic Headache and Type II Whiplash Associated Disorder: a Multi-center Randomized Clinical Trial
Brief Title: Manipulation and Dry Needling in Patients With Cervicogenic Headache and WAD II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, PhD, DPT, FAAOMPT, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT0018
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Cervicogenic Headache; Whiplash Injuries
Keywords: Headache; Whiplash
MeSH Terms: conditions — Post-Traumatic Headache; Whiplash Injuries; Headache | interventions — Dry Needling; Manipulation, Spinal; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry Needling,Thrust Manipulation (Experimental): Dry needling to the craniofacial, upper cervical, and cervicothoracic regions. High-velocity thrust manipulation to the upper cervical spine, mid/lower cervical spine, and cervicothoracic spinal regions.
  Interventions: Other: Dry Needling,Thrust Manipulation
- Exercise,Non-thrust Mobilization (Active Comparator): Nonthrust joint mobilization to the upper cervical spine, mid/lower cervical spine, and cervicothoracic spinal regions. Cranio-cervical flexion exercises, peri-scapular progressive resistance exercises, and electrothermal modalities
  Interventions: Other: Exercise,Non-thrust Mobilization

INTERVENTIONS:
Other: Dry Needling,Thrust Manipulation — HVLA thrust manipulation to upper cervical and upper thoracic regions. Dry needling to cervicothoracic and craniofacial regions. Up to 8 treatment sessions over 4 weeks.
  Other Names: Spinal Manipulation; Dry Needling
  Arms: Dry Needling,Thrust Manipulation
Other: Exercise,Non-thrust Mobilization — Non-thrust mobilization and exercise to upper cervical and upper thoracic regions. Up to 8 treatment sessions over 4 weeks.
  Other Names: Exercise; Non-thrust Mobilization
  Arms: Exercise,Non-thrust Mobilization

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with cervicogenic headaches associated with type II whiplash associated disorder: non-thrust mobilization and exercise versus thrust manipulation and dry needling. Physical therapists commonly use all of these techniques to treat cervicogenic headaches. This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patients with cervicogenic headaches and type II whiplash associated disorder will be randomized to receive 1-2 treatment sessions per week for 4 weeks (up to 8 sessions total) of either: (1) dry needling and upper cervical high-velocity low-amplitude thrust manipulation, or (2) exercise and non-thrust mobilization.

ELIGIBILITY:
Inclusion Criteria:

1. Subacute (> 4 weeks) or chronic type II whiplash associated disorder. Neck pain and headache following motor vehicle accident with reduced range of motion & point tenderness.
2. Diagnosis of cervicogenic headache as defined by Cervicogenic Headache International Study Group criteria.
3. Headache frequency of at least one per week since the whiplash injury.
4. Headache intensity of greater than 2/10 on the NPRS.
5. Neck pain intensity of greater than 2/10 on the NPRS.
6. Neck Disability Index score of greater than 10/50 on the NDI.

Exclusion Criteria:

1. WAD I (neck pain, but no physical signs), WAD III (neck pain and neurological signs), WAD IV (neck pain + fracture/dislocation).
2. Positive screen for cervical radiography (Canadian C-Spine Rules).
3. Bilateral headaches (typical of tension type headaches).
4. Diagnosis / signs & symptoms of concussion (confusion, disorientation, or impaired consciousness; loss of memory for events immediately before or after the MVA; and one or more of the following: nausea, vomiting, visual disturbances, vertigo, gait and/or postural imbalance, and impaired memory and/or concentration).
5. Diagnosis of fibromyalgia.
6. Presence of any of the following atherosclerotic risk factors: hypertension, diabetes, heart disease, stroke, transient ischemic attack, peripheral vascular disease, smoking, hypercholesterolemia, or hyperlipidemia.
7. Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e., tumor, fracture, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, etc.).
8. Diagnosis of cervical spinal stenosis.
9. Bilateral upper extremity symptoms.
10. Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes).
11. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

    1. Muscle weakness involving a major muscle group of the upper extremity.
    2. Diminished upper extremity deep tendon reflex of the biceps, brachioradialis, triceps or superficial flexors
    3. Diminished or absent sensation to pinprick in any UE dermatome.
12. Prior surgery to the head, neck, or thoracic spine.
13. Physical therapy or chiropractic treatment for neck pain and/or headache in the past 3 months.
14. Any condition that might contraindicate spinal manipulative therapy or dry needling.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Headache Intensity (Numeric Pain Rating Scale, 0-10) (Rating Score) | Baseline, 4 weeks, 3 months, 6 months
  Rating Score on 0-10 scale. Baseline score must exceed 2/10 to be included. Lower scores indicate less pain intensity.
  the study.

SECONDARY OUTCOMES:
Change in Global Rating of Change Score for Headaches | 6 months
  Rating score for self perceived change with range of -7 to +7. Higher scores indicate greater improvement.
Change in Global Rating of Change Score for Neck Pain | 6 months
  Rating score for self perceived change with range of -7 to +7. Higher scores indicate greater improvement.
Change in Medication Intake (Frequency of medication intake in last week) | Baseline, 6 months
  Over the counter and prescription medication
Change in Headache Duration (Total hours of headaches in the last week) | Baseline, 4 weeks, 3 months, 6 months
  Total hours of headaches in the last week
Change in Headache Frequency (Number of headaches in the last week) | Baseline, 4 weeks, 3 months, 6 months
  Number of headaches in the last week
Change in Disability (Neck Disability Index, 0-50 points) | Baseline, 4 weeks, 3 months, 6 months
  10 Questions each worth 0-5 points with maximum score of 50 points possible. Lower scores indicate lower disability levels. Baseline score must exceed 10/50 to be included in study.
Change in Neck Pain Intensity (Numeric Pain Rating Scale, 0-10 points) | Baseline, 4 weeks, 3 months, 6 months
  Rating score 0-10 points. Lower scores indicate lower pain intensity. Baseline score must exceed 2/10 to be included
Change in Pain Catastrophizing Scale (0-52 points) | Baseline, 6 months
  13 questions each worth 0-4 points with maximum score of 52 points. Lower scores indicate less pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, PhD, DPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Alabama Physical Therapy & Acupuncture, Montgomery, Alabama, United States

IPD SHARING:
Plan to Share IPD: No